CLINICAL TRIAL: NCT05342142
Title: Effects of 12-week Aerobic and Resistance Exercises on Alexithymia, Depression and Quality of Life in Geriatric Individuals
Brief Title: Effects of 12-week Exercises on Alexithymia, Depression and Quality of Life in Geriatric Individuals
Acronym: EXQUALITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EXQUALITY
Record Dates: First submitted 2022-04-12; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Depression; Alexithymia; Quality of Life; Physical Inactivity
Keywords: Depression; Alexithymia; Quality of Life; Elderly; Exercise
MeSH Terms: conditions — Depression; Affective Symptoms; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): Exercise program consisting of 12 weeks of aerobic and resistance exercises
  Interventions: Behavioral: Aerobic and ResistanceExercise
- Control (No Intervention): No intervention will be made

INTERVENTIONS:
Behavioral: Aerobic and ResistanceExercise — Exercise program consisting of 12 weeks of aerobic and resistance exercises
  Arms: Exercise

SUMMARY:
The aim of this study is to investigate the effects of aerobic and resistance exercises on depression, alexithymia levels and quality of life of elderly individuals.

DETAILED DESCRIPTION:
In this study, investigators hypothesized that aerobic and resistance exercises can increase the quality of life of elderly individuals by reducing their depression and alexithymia levels. The aim of this study is to investigate the effects of aerobic and resistance exercises on depression, alexithymia levels and quality of life of elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over who volunteered to participate in the study,
* Conscious and without communication problems,
* No orthopedic injury that prevents walking
* Those who are physically inactive according to the International Physical Activity Assessment Questionnaire
* Those who have sufficient motivation to participate in the exercise program (will be evaluated by a one-on-one interview by the researchers)
* Being eligible to participate in an exercise program after a cardiac examination (resting ECG and questioning of cardiac symptoms, advanced tests such as exercise ECG test if necessary) performed by the physician.

Exclusion Criteria:

* Having a history of neuromuscular disease
* Serious medical condition (eg advanced malignancy or major neurological, psychiatric or endocrine disease, respiratory failure, etc.) that would prevent the person from participating in exercise training.
* Less than 1 year life expectancy
* Having an orthopedic injury that prevents walking
* Presence of advanced sensory deficit
* Having visual and hearing problems
* Not having sufficient communication skills (Mini Mental Test score below 24 points)
* Not having agreed to participate in the study
* Uncontrolled hypertension
* Not being found suitable for exercise in the examination performed by physicians and physiotherapists

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — 65 years and over
Enrollment: 70 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Depression | 1 week
  depression level as measured by the geriatric depression scale (min:0, max:15, 5 or more means more depression)
Alexythimia | 1 week
  Alexythimia level as measured by the toronto Alexythimia scale (min:0, max:100, 61 ore more means more alexythimia)
quality of life | 1 week
  level of quality of life measured by health related quality of life scale(min:24, max:120, high levels means low quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Training And Research Hospital
Locations (1):
- Sultan Abdülhamid Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No